CLINICAL TRIAL: NCT01560312
Title: Renal Denervation - Hope for Patients With Refractory Hypertension?
Brief Title: Renal Denervation in Refractory Hypertension
Acronym: PRAGUE-15
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on analysis of our data after the Symplicity-3 trial announcement, decision for study termination was done.
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other); University Hospital Olomouc (Other); Cardiocenter Podlesí, Trinec, Czech Republic (Unknown)
Responsible Party: Principal Investigator, Petr Widimsky, MD, Head of Cardiocenter, 3rd Faculty of Medicine, Charles University, Czech Republic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Charles University
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Hypertension; Resistant to Conventional Therapy
Keywords: Renal denervation; Resistant hypertension; Spironolactone; Long-term Outcome
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal denervation (Experimental): Renal denervation (Symplicity® Catheter System™) + conventional antihypertensive medical treatment without spironolactone (spironolactone can be taken only if started before randomization)
  Interventions: Device: Renal denervation (Symplicity® Catheter System™)
- Medical treatment (No Intervention): Conventional antihypertensive treatment including spironolactone (if not contraindicated).
  One year after randomization, renal denervation can be performed according to the physician's decision based on the BP levels and if patient desires the procedure.

INTERVENTIONS:
Device: Renal denervation (Symplicity® Catheter System™) — 4-6 ablation in both renal arteries using the Symplicity® Catheter System™ (Ardian/Medtronic)
  Arms: Renal denervation

SUMMARY:
Open, multicenter, randomized study is enrolling patients in 3 sites in Czech Republic. Patients with refractory hypertension will be randomized in 1:1 manner either to renal denervation plus optimal medical antihypertensive treatment without spironolactone or to antihypertensive treatment alone including spironolactone if not contraindicated. The primary end-point is change in Systolic and Diastolic Blood Pressure (BP) between baseline and 1 year after randomization evaluated by 24-hours BP monitoring. Expected enrollment is 120 patients. Patients follow-up is planned for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Refractory hypertension with office SBP > 140 mmHg
* SBP > 130 during 24-hours Holter blood pressure monitoring
* Treatment with the least 3 antihypertensive medications including diuretics in optimal doses
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Secondary forms of hypertension
* Chronic renal disease (serum creatinine > 200 umol/l)
* Pregnancy
* History of myocardial infarction or stroke in last 6 months
* Severe valvular stenotic disease
* Anatomic abnormalities and variants of renal artery including aneurysms, severe stenosis, reference diameter < 4 mm or length < 20 mm
* Increased bleeding risk (thrombocytopenia < 50, INR > 1.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure difference | 6 months
  Systolic and Diastolic blood pressure difference between baseline and 6 months post-randomization. Blood pressure will be evaluated using 24-hours monitoring.

SECONDARY OUTCOMES:
Blood pressure differences similar to primary outcome | 1 year, 2 years, 3 years
  Systolic and Diastolic BP differences (comparison between baseline and evaluated time period) will be measured using 24-hours monitoring and also at office.
Change of blood laboratory parameters and renal function | 6 months, 1, 2, 3 years
  changes in blood concentrations of renin, aldosterone, metanephrines and renal function
Post-denervation renal anatomy assessment | 1 year
  CT angiography will be performed 1 year after RDN

CONTACTS AND LOCATIONS:
Overall Officials: Petr Widimsky, Prof, MD, Principal Investigator — Charles University, Prague, Czech Republic; Jiri Widimsky, Prof.MD., Principal Investigator — General University Hospital
Locations (3):
- Czechia (3):
  - Cardiocenter, University Hospital Olomouc, Olomouc
  - Jiri Widimsky, Prague
  - Cardiocenter Podlesi, Třinec